CLINICAL TRIAL: NCT02924012
Title: Energy Demand in a Video Game Active Session and Potencial to Promove Post Exercise Hypotension in Hypertensive Women
Brief Title: Active Video Game and Potential to Cause Post-exercise Hypotension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Taís Feitosa da Silva, Master, Federal University of Paraíba
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VGA-HYP
Record Dates: First submitted 2016-10-03; First posted 2016-10-05 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-09

CONDITIONS: Hypertension
Keywords: post exercise hypotension; exercise; video games
MeSH Terms: conditions — Hypertension; Post-Exercise Hypotension; Motor Activity | interventions — Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- active video game (Experimental): An active game session lasting 40 minutes
  Interventions: Other: video game active
- sedentary video game (Other): An sedentary game session lasting 40 minutes
  Interventions: Other: sedentary video game
- walking (Other): An walking lasting 40 minutes
  Interventions: Other: walking

INTERVENTIONS:
Other: video game active — The session lasted 40 minutes. The participants held an active video game session. At the end they were monitored for 60 minutes at rest.
  Other Names: AVG
  Arms: active video game
Other: sedentary video game — The session lasted 40 minutes. The participants held an sedentary video game session, using the traditional joystick. At the end they were monitored for 60 minutes at rest.
  Other Names: SVG
  Arms: sedentary video game
Other: walking — The session lasted 40 minutes. The participants held a walk using the treadmill. At the end they were monitored for 60 minutes at rest.
  Other Names: WAL
  Arms: walking

SUMMARY:
The aim of this study was to determine the energy demand and the potential to promote reduce blood pressure of an active video game (AVG). Fourteen hypertensive (56.4 ± 7.5 years) held a session AVG and traditional sedentary video game sessions (SVG) and walk (WAL), as negative and positive controls, in order determined randomly. During the sessions, they were observed oxygen consumption and energy expenditure (EE). Blood pressure (BP) and cardiac autonomic modulation (CAM) were measured at rest and every 15 minutes of a 60 minute period of recovery activities. It was also applied a rating scale of pleasure (enjoyment scale).

DETAILED DESCRIPTION:
Volunteers: In a previous pilot study, seven women who had systolic blood pressure (SBP) of resting 128.9 ± 9.4 mmHg obtained a reduction to 116.9 ± 7.0 mmHg 60 minutes after a workout with AVG. These data resulted in an effect size of 1.05. Adopting an α error of 0.05 and statistical power of 0.95, estimated a minimum sample size of 12 volunteers. effectively participated in the study 14 hypertensive women aged between 47 and 68 years (56.4 ± 7.5 years). In addition to the diagnosis of hypertension, they should perform with pressure values of at least 130/90 mmHg and no greater than 160/110 mmHg in measurements made in the days before the study and on the day of data collection. They should still be postmenopausal women, being overweight or obesity grade I (BMI between 25 and 34.9 kg / m2), not be practicing systematic physical exercise for at least three months and not be suffering from labyrinthitis. They would be excluded from the study volunteers who initiate any antihypertensive treatment during the study period, presented difficulties to perform the AVG games or take him more than four weeks to complete all experimental procedures.

The research project was approved by the Research Ethics Committee of the Health Science Center - UFPB under the nº0621 / 14 protocol. After informed about all the procedures, the volunteers signed a Consent and Informed (IC) according to the resolution 466/12 of the National Health Council of Brazil.

Study design: the volunteers held an AVG session, an internal control session composed of sedentary video game (SVG) and an external control session consists of a walking exercise (WAL) with a minimum of 48 hours between sessions and order determined randomly. In all sessions, during activities, they were instrumented with portable gas analyzer for measuring energy expenditure (EE) accelerometer to quantify performed movements and heart rate monitor to evaluate the behavior of heart rate (HR). Blood pressure measurements (BP) and cardiac autonomic modulation (CAM) were performed at rest and every 15 minutes a period 60 minutes of recovery activities. In these same times it was applied a rating scale of pleasure in activities (enjoyment scale) (Figure 1).

Pre experimental procedures: prior to the experimental sessions, blood pressure measurements, physical activity and blood collection were made to characterize the participants. Personal information on the drugs used and collected and they were given a list containing rich foods and medicines caffeine could not be ingested 24 before each experimental session.

Adaptation activities: the participants underwent three sessions of adaptation and learning the handling of active and sedentary games and walking on a treadmill. The sessions lasted 10 to 40 minutes, with an interval of 48 hours between sessions and at least 72 hours between the last session of adaptation and the first test session. The intensity adopted in these sessions was free, but participants were encouraged to achieve moderate intensity on the treadmill exercise (60% to 85% of maximum heart rate). They were also taught to respond to the subjective perception questionnaires effort and enjoyment scale.

Video active game: the console was the Xbox 360 with Kinect sensor (Foxconn®, New Taipei, China) and the game used was Dance Central (Harmonix Music Systems - Microsoft Games Studios). The difficulty level of the game was adopted the beginner, since the participants had no previous experience with AVG. In the game used, bodily movements are similar to dance steps with the use of different songs from pop style referring to the 1970, 1980, 1990 and 2000. The session lasted 40 minutes.

Video game sedentary: we used the Dance Dance Revolution® (SSD Company Ltd., Shiga, Japan) for Playstation 2® (San Mateo, CA, USA), where the practitioner simulated synchronized dances of similar songs to those used in gyms, however using the joystick traditionally known, so that remained seated throughout the session. The duration of the game was 40 minutes.

walking exercise: the participants performed a walking session on a treadmill (Moviment, Brudden Ltda, São Paulo, Brazil) lasting 40 minutes and previously prescribed intensity between 60% and 80% of maximum heart rate.

Accelerometry: an accelerometer used was brand Actigraph® GT3 X (Pensacola, USA) for evaluating the acceleration of the body, calibrated according to the manufacturer's specifications. The adopted time interval was 60 seconds and output data expressed as mean counts per minute. The unit was set at waist height, the right hand by a strap of elastic and adjustable buckle. At the end of the records, data were transferred to a computer and analyzed using the SAS 9.2 software (SAS Institute Inc., Cary, NC 25513). The adopted referêcia values were 0-99 counts / min-1, considered sedentary activity, 100-1951 counts / min-1, light activity, 1952-5724 counts / min-1 was moderate activity and from 5725 counts / min-1, seen vigorous activity, according Freedson et al (113) Energy demand: it was made by gas analysis through the analyzer portable lung gases K4b2 (Cosmed Copyritgh ©, Rome, Italy) validated the study by McLaughlin et al (114). This equipment enables verification in each breath, respiratory parameters, measuring the oxygen consumption (VO2) and carbon dioxide production during exercise. The device was calibrated according to the manufacturer's recommendations. The variables measured by this instrument were the DE and VO2. The measurements were performed at rest (for five minutes) and during experimental sessions.

Heart rate and perceived exertion: HR was measured using a heart rate monitor brand Polar RS800CX model (Polar ElectroOy, Kempele, Finland). The measurements were made after 10 minutes at rest and every 5 minutes Durantes exercises. In the same times that HR was measured, the Subjective Perception Scale of Borg effort (Noble and Borg et al, 1983), with scale 6-20 points, was presented to the participants and asked who said they had their feelings of stress.

Enjoyment Scale: This scale has been validated for use in the adult population according to Graves et al. (2008). It consists of 18 items that assessed the level of pleasure / enjoyment from levels ranging from "I like" to "I hate" in that the higher the sum of these points, pleasure / enjoyment the activity performed provided. This scale was presented to participants at the beginning of each study session and the same to answer the end of each study session.

Blood pressure: before the start of each session, participants were asked to stay 15 minutes at rest and sitting. After this period was found resting BP. Further measures were taken immediately at the end of the experimental session and every 15 minutes during a 60-minute recovery period, the volunteers seated throughout this period. These measurements were performed by the oscillometric method with the use of ambulatory monitoring apparatus PA (DYNAMAPA) following the V Brazilian Guidelines on BP ambulatory monitoring (ABPM) (ALESSI, A; BRANDÃO, A.;. PIERIN et al, 2005). three pressure taps were made for each measure and considered the two closest values.

Cardiac Autonomic Modulation (CAM): Immediately after each measurement of BP, we evaluated the MAC through the HR variability, using a monitor brand Polar RS800CX (PolarElectroOy, Kempele, Finland). The volunteers were seated and the record was made for a minimum of 10 minutes. Data were transferred to a computer provided with software of the same manufacturer and then transferred to the Kubios HRV software, version 2.0 (University of Kuopio, Finland). Data were analyzed in the time domain, being considered the average (RRM) and the standard deviation of the individual intervals RR (SDNN), the root mean square of successive differences between adjacent RR (RMSSD) and the percentage of successive differences between RR intervals greater than 50 ms (pNN50). In the frequency domain, they were considered low frequency bands (0:04 to 00:15 Hz) (LF) and high frequency (0.15 to 0.4 Hz) (AF). It was also adopted the low ratio frequency / high frequency as sympathetic-vagal balance (LF / HF).

Statistical analysis: Data are mean and standard error of the mean. the Shapiro-Wilk tests were used to verify the normality and Levene to check homogeneity. One-way ANOVA was used to compare the resting values. For comparisons between measurements during and after the experimental sessions, it adopted the two-way ANOVA test. Data were analyzed using the GraphPad Prism 6.0 software (GraphPad, San Diego, CA, USA), a significance of p <0.05.

ELIGIBILITY:
Inclusion Criteria:

Hypertension Diagnosis Be postmenopausal Display overweight or obesity grade I (BMI between 25 and 34.9 kg / m2) Not practicing systematic physical exercise for at least three months Not carry labyrinthitis

Exclusion Criteria:

Start any antihypertensive treatment during the study period Have difficulty to perform the AVG games Take more than four weeks to complete all experimental procedures

Ages: 47 Years to 68 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-05; Primary Completion 2015-08 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | Sixty minutes after AVG, SVG or WAL
  Before the Start All such sessions, as requested Participants Were one Stay 15 Minutes Resting and sitting. After this period was checked PA Home. New Outlets Were measures immediately At the end of the session and experimental one every 15 minutes during hum 60 Minutes Recovery Period, with as sitting voluntary period During this ALL. These measures Were performed hair oscillometric method with the use of ambulatory monitoring apparatus PA (DYNAMAPA) following the V Brazilian Guidelines on BP ambulatory monitoring (ABPM) (ALESSI, A; BRANDÃO, A. ;. PIERIN et al, 2005). Were Made Three pressure sockets one measure and considered each The two values Closer.

SECONDARY OUTCOMES:
Quantifying the movements | Forty minutes duration AVG, SVG or WAL
  It used an accelerometer brand Actigraph® GT3 X (Pensacola, USA) for evaluating the acceleration of the body, calibrated according to the manufacturer's specifications. The adopted time interval was 60 seconds and output data expressed as mean counts per minute. The unit was set at waist height, the right hand by a strap of elastic and adjustable buckle. At the end of the records, data were transferred to a computer and analyzed using the SAS 9.2 software (SAS Institute Inc., Cary, NC 25513). The adopted referêcia values were 0-99 counts / min-1, considered sedentary activity, 100-1951 counts / min-1, light activity, 1952-5724 counts / min-1 was moderate activity and from 5725 counts / min-1, seen vigorous activity, according Freedson et al
Cardiac autonomic modulation | Sixty minutes after AVG, SVG or WAL
  Immediately after each measurement of BP was assessed by MAC HR variability, using a monitor label Polar RS800CX (PolarElectroOy, Kempele, Finland). The volunteers were seated and the record was made for a minimum of 10 minutes. Data were transferred to a computer provided with software of the same manufacturer and then transferred to the Kubios HRV software, version 2.0 (University of Kuopio, Finland). Data were analyzed in the time domain, being considered the average (RRM) and the standard deviation of the individual intervals RR (SDNN), the root mean square of successive differences between adjacent RR (RMSSD) and the percentage of successive differences between RR intervals greater than 50 ms (pNN50). In the frequency domain, they were considered low frequency bands (0:04 to 00:15 Hz) (LF) and high frequency (0.15 to 0.4 Hz) (AF). It was also adopted the low ratio frequency / high frequency as sympathetic-vagal balance (LF / HF).
Enjoyment scale | Sixty minutes after AVG, SVG or WAL
  This scale has been validated for use in the adult population according to Graves et al. (2008). It consists of 18 items that assessed the level of pleasure / enjoyment from levels ranging from "I like" to "I hate" in that the higher the sum of these points, pleasure / enjoyment the activity performed provided. This scale was presented to participants at the beginning of each study session and the same to answer the end of each study session.
Energy expenditure | Forty minutes duration AVG, SVG or WAL
  Was made by gas analysis through the analyzer portable lung gases K4b2 (Cosmed Copyritgh ©, Rome, Italy) validated the study by McLaughlin et al. This equipment enables verification in each breath, respiratory parameters, measuring the oxygen consumption (VO2) and carbon dioxide production during exercise

IPD SHARING:
Plan to Share IPD: No